CLINICAL TRIAL: NCT00923117
Title: A Phase II Trial of Sunitinib in the Treatment of Recurrent Malignant Gliomas
Brief Title: Sunitinib to Treat Recurrent Brain Cancer
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: The study was terminated based on results of an interim analysis for futility.
Sponsor: National Cancer Institute (NCI) (NIH)
Responsible Party: Principal Investigator, Teri Kreisl, M.D., Principal Investigator, National Institutes of Health Clinical Center (CC)
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 080168; 08-C-0168; NCT00713388 (obsolete NCT alias)
Record Dates: First submitted 2009-06-17; First posted 2009-06-18 (Estimated); Results first posted 2013-06-25 (Estimated); Last update posted 2015-09-30 (Estimated); Status verified 2014-07

CONDITIONS: Glioblastoma Multiforme; Malignant Gliomas; Anaplastic Gliomas
Keywords: Glioblastoma; Chemotherapy; Anti-Angiogenesis; Radiation; Brain Tumor; Malignant Glioma; Glioblastoma Multiforme
MeSH Terms: conditions — Glioblastoma; Glioma; Brain Neoplasms | interventions — Sunitinib

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Bevacizumab resistant patients (Experimental): Patients who had tumor progression while treated with bevacizumab.
  Interventions: Drug: Sutent (sunitinib)
- Bevacizumab naive patients (Experimental): Patients with progressive tumor who have not been treated with bevacizumab.
  Interventions: Drug: Sutent (sunitinib)

INTERVENTIONS:
Drug: Sutent (sunitinib) — Oral dose 37.5 mg daily on a continuous 4 week cycle

SUMMARY:
Background:

One way tumors are able to grow is by forming new blood vessels that supply them with nutrients and oxygen.

Sunitinib blocks certain proteins on the surface of tumor and blood vessel cells that are involved with the formation of new blood vessels.

Blocking these proteins may prevent the tumor cells or blood vessels from continuing to grow.

Objectives:

To determine whether sunitinib can cause tumors to shrink or stabilize in patients with recurrent brain cancer.

Eligibility:

Patients 18 years of age or older with brain cancer whose disease has worsened after standard treatment with surgery, radiation.

Design:

Patients take a sunitinib pill once a day in 4-week treatment cycles. Treatment may continue as long as the tumor remains stable or decreases in size and the side effects of treatment are tolerated.

Routine blood tests are done every 2 weeks during the first 8 weeks of treatment and then every 4 weeks after that.

Magnetic resonance imaging (MRI) scans are done before starting treatment (at baseline) and at the end of every 4-week cycle to monitor tumor growth.

Positron emission tomography (PET) scans are done at baseline and at the end of the first cycle.

Neurological and physical examinations are done at baseline, at week 2 of treatment and at the end of every treatment cycle.

Health-related quality of life is assessed every 4 weeks.

Pregnancy tests, electrocardiograms and echocardiograms are repeated as needed.

DETAILED DESCRIPTION:
Background:

Solid tumors have multiple mechanisms for stimulating angiogenesis with the vascular endothelial growth factor (VEGF)-kinase insert domain receptor (KDR) axis being only one of them. Sunitinib, through its multiple tyrosine kinase receptor targets, represents an attempt to capitalize on the concept of targeting multiple mechanisms responsible for glioma-associated angiogenesis. Sunitinib inhibits platelet derived growth factor receptor (PDGFR) and c-kit (stem cell factor (SCF) receptor) at nanomolar concentrations. The combination blocks all three known major glioma-mediated angiogenic mechanisms (VEGF, c-kit, PDGF). Based on this scientific rationale, the promising anti-glioma activity of sunitinib in preclinical models, and the promising clinical data in patients with gliomas treated with other VEGF inhibitors, we are now proposing a phase II trial of sunitinib in patients with recurrent malignant gliomas.

Objectives:

To evaluate the anti-glioma activity of sunitinib in patients with recurrent malignant gliomas who are either naive or resistant to prior bevacizumab therapy.

Eligibility:

Patients with recurrent malignant glioma are eligible for this study.

Design:

This is a phase II study with a target enrollment of 64 (32 with glioblastoma multiforme (GBM) and 32 with anaplastic glioma (AG)) patients who have not progressed on prior treatment with anti-VEGF therapy, and 64 (32 with GBM and 32 with AG)patients who have progressed on prior bevacizumab therapy.

Sunitinib will be self-administered orally at 37.5 mg daily, with dose adjustments allowed for toxicity and concomitant drug interactions.

The primary endpoint is six-month progression free survival for both arms of the study.

We performed an interim analysis (see below) and after consulting with the pharmaceutical company (Pfizer) we believe that ending the study is the most appropriate course of action to take.

In the original design of the trial, for the AG stratum, the agent will be considered effective if at least 14 patients have not progressed by 6 months. Now, we have observed one out 10 Bev-naïve who haven't progressed by 6 months. Then given one patient in the first 10 patients whose PFS >=6, the conditional probability of observing at least 14 out of 32 patients who are 6 month-PFS is only 43% even if the true 6 months-PFS is 55%. Since in the first 10 patients, we only observed one patient with PFS>=6 months, it is unlikely that the true 6 month-PFS is 55%. The conditional power would be close to zero, if the true 6 month-PFS close to 10% as observed so far. Based on the conditional probability, the chance of a positive study is small, and hence the trial should be considered stopped for futility.

For Bev-resistant patients, because in the first 12 patients none had PFS >= 6 months the conditional probability of declaring the agent being effective is even lower and equals 12%, if the true PFS at 6 months is 55%. Essentially there is little chance that the agent can be declared effective.

ELIGIBILITY:
* INCLUSION CRITERIA:

  1. Patients with histologically proven intracranial malignant glioma will be eligible for this protocol. Malignant gliomas include glioblastoma multiforme (GBM), gliosarcoma (GS), anaplastic astrocytoma (AA), anaplastic oligodendroglioma (AO), anaplastic mixed oligoastrocytoma (AMO), or malignant astrocytoma NOS (not otherwise specified).
  2. Patients may have received prior therapy with bevacizumab, but not within six weeks of starting treatment with sunitinib. Patients who received prior therapy with bevacizumab must have demonstrated radiographic disease progression while being treated with bevacizumab.
  3. Patients must have progressed after radiation and temozolomide therapy and have an interval of greater than or equal to 4 weeks from the completion of radiation therapy to study entry. If the patient has had prior stereotactic radio surgery, true tumor progression must be corroborated by fludeoxyglucose 18F (FDG)-positron emission tomography (PET) or magnetic resonance (MR) spectroscopy imaging.
  4. Patients must have evidence of tumor progression by contrast enhanced perfusion magnetic resonance imaging (MRI) or computed tomography (CT) scan. This scan should be performed within 14 days prior to registration and on a five-day stable dose of steroids. If the steroid dose is increased between the date of imaging and registration, a new baseline MR/CT is required. The same type of scan (i.e., MRI or CT) must be used throughout the period of protocol treatment for tumor measurement.
  5. Patients having undergone recent resection of recurrent or progressive tumor will be eligible as long as all of the following conditions apply:
* They have recovered from the effects of surgery.
* Residual disease following resection of recurrent tumor is not mandated for eligibility into the study. To best assess the extent of residual disease post-operatively, a CT/MRI should be done:

  * no later than 96 hours in the immediate post-operative period, or
  * at least 4 weeks post-operatively, and
  * within 14 days of registration, and
  * on a steroid dosage that has been stable for at least 5 days.

    f) Normal organ and marrow function defined as: total leukocyte count greater than or equal to 3000 cells/ul, absolute neutrophil count (ANC) greater than or equal to 1500 cells/ul, platelet count greater than or equal to 100,000 cells/ul, serum creatinine less than or equal to 2.0 times the upper limit of normal, and bilirubin less than or equal to 1.5 times the upper limit of normal, hemoglobin greater than or equal to 9.0 g/dL , serum calcium less than or equal to 12.0 mg/dL, aspartate aminotransferase (AST)/alanine aminotransferase (ALT) less than or equal to 1.5 times the upper limit of normal, prothrombin time (PT) less than or equal to 1.5 upper limits of normal (ULN). Eligibility level for hemoglobin may be reached by transfusion.

    g) The effects of sunitinib on the developing human fetus at the recommended therapeutic dose are unknown. Women of child-bearing potential and men must agree to use adequate contraception (hormonal or barrier method of birth control; abstinence) prior to study entry and for the duration of study participation. Should a woman become pregnant or suspect she is pregnant while participating in this study, she should inform her treating physician immediately.

    h) All patients or their previously designated durable power of attorney (DPA) (if the patient is deemed by the treating physician to be impaired or questionably impaired in such a way that the ability of the patient to give informed consent is questionable) must sign an informed consent indicating that they are aware of the investigational nature of this study.

    i) Patients must be greater than or equal to 18 years old, and with a life expectancy greater than 8 weeks.

    j) Patients must have a Karnofsky performance status of greater than or equal to 60.

    k) Patients must have recovered from the toxic effects of prior therapy: 2 weeks from any investigational agent, two weeks from vincristine, 6 weeks from nitrosoureas, 3 weeks from procarbazine, 1 week for non-cytotoxic agents, (e.g., interferon, tamoxifen, thalidomide, cis-retinoic acid, etc.), and 4 weeks from other cytotoxic therapy. Any questions related to the definition of non-cytotoxic agents should be directed to the Study Chair.

    l) Patients must not have any significant medical illnesses that in the investigator's opinion cannot be adequately controlled with appropriate therapy or would compromise the patients' ability to tolerate this therapy.

    m) This study was designed to include women and minorities, but was not designed to measure differences of intervention effects. Males and females will be recruited with no preference to gender. No exclusion to this study will be based on race. Minorities will actively be recruited to participate.

EXCLUSION CRITERIA:

1. Patients who, in the view of the treating physician, have significant active cardiac, hepatic, renal, or psychiatric diseases are ineligible.
2. Patients with a history of prior therapy directed against vascular endothelial growth factor (VEGF) (e.g. sorafenib, pazopanib, Zactima (ZD6474), AZD2171), with the exception of bevacizumab, will not be allowed to enroll.
3. Concurrent use of other standard chemotherapeutics or investigative agents.
4. Patients known to have a malignancy (other than their malignant glioma) that has required treatment in the last 12 months and/or are expected to require treatment in the next 12 months (except non-melanoma skin cancer or carcinoma in-situ in the cervix).
5. Patients who have an active infection.
6. Pregnant (positive pregnancy test) or nursing women. Both fertile men and women must agree to use adequate contraceptive measures during study therapy and for at least 3 months after the completion of sunitinib therapy.
7. Concurrent anti-coagulation or anti-platelet medication (including aspirin, non-steroidal anti-inflammatory agents, cyclooxygenase -2 (COX-2) inhibitors).
8. Serious or non-healing wound, ulcer or bone fracture
9. History of any of the following within 6 months of study entry: abdominal fistula, gastrointestinal perforation, intra-abdominal abscess, stroke, myocardial infarction or unstable angina. Patients will not undergo diagnostic screening for any of these conditions.
10. Invasive procedures defined as follows:

    * Major surgical procedure, open biopsy or significant traumatic injury within 28 days prior to Day 1 therapy
    * Anticipation of need for major surgical procedures during the course of the study
    * Core biopsy within 7 days prior to start of therapy
11. Uncontrolled hypertension (greater than 150/100 mmHg) while on antihypertensive medications.
12. New York Heart Association class II or greater congestive heart failure.
13. Serious cardiac arrhythmia requiring medication.
14. Evidence of bleeding diathesis, coagulopathy, or international normalized ratio (INR) greater than 1.5.
15. History of allergic reactions attributed to compounds of similar chemical or biologic composition to sunitinib.
16. Patients receiving any enzyme inducing anti-epileptic drugs (EIAEDs) and other potent cytochrome P450 3A4 (CYP3A4) modulators (per Appendixes B and C) within two weeks prior to treatment start are ineligible.
17. Baseline echocardiogram with ejection fraction less than 50% or greater than or equal to 20% decrease from a prior study
18. corrected QT interval(QTc) interval greater than 500 msec on baseline electrocardiogram (EKG).
19. Human immunodeficiency virus (HIV)-positive patients on combination antiretroviral therapy are ineligible because of the potential for pharmacokinetic interactions with sunitinib.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 87 (Actual)
Dates: Start 2008-06; Primary Completion 2012-06 (Actual); Study Completion 2012-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Teri N Kreisl, M.D., Principal Investigator — National Cancer Institute (NCI)
Locations (1):
- National Institutes of Health Clinical Center, 9000 Rockville Pike, Bethesda, Maryland, United States

REFERENCES:
- [Background] Jemal A, Siegel R, Ward E, Murray T, Xu J, Thun MJ. Cancer statistics, 2007. CA Cancer J Clin. 2007 Jan-Feb;57(1):43-66. doi: 10.3322/canjclin.57.1.43. PMID 17237035
- [Background] Prados MD, Schold SC Jr, Fine HA, Jaeckle K, Hochberg F, Mechtler L, Fetell MR, Phuphanich S, Feun L, Janus TJ, Ford K, Graney W. A randomized, double-blind, placebo-controlled, phase 2 study of RMP-7 in combination with carboplatin administered intravenously for the treatment of recurrent malignant glioma. Neuro Oncol. 2003 Apr;5(2):96-103. doi: 10.1093/neuonc/5.2.96. PMID 12672281
- [Background] Prados MD, Warnick RE, Mack EE, Chandler KL, Rabbitt J, Page M, Malec M. Intravenous carboplatin for recurrent gliomas. A dose-escalating phase II trial. Am J Clin Oncol. 1996 Dec;19(6):609-12. doi: 10.1097/00000421-199612000-00016. PMID 8931682
- See also: NIH Clinical Center Detailed Web Page — http://clinicalstudies.info.nih.gov/cgi/detail.cgi?B_2008-C-0168.html

RESULTS

PARTICIPANT FLOW:
Groups:
- Bevacizumab Resistant Patients: Patients who had tumor progression while treated with bevacizumab. Oral dose Sutent (sunitinib) 37.5 mg daily on a continuous 4 week cycle.
- Bevacizumab Naive Patients: Patients with progressive tumor who have not been treated with bevacizumab.Oral dose Sutent (sunitinib) 37.5 mg daily on a continuous 4 week cycle.
Period: Overall Study
Arm/Group | Bevacizumab Resistant Patients | Bevacizumab Naive Patients
Started | 44 | 43
Completed | 44 | 43
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Bevacizumab Resistant Patients | Bevacizumab Naive Patients | Total
Number analyzed (Participants) | 44 | 43 | 87
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 37 | 39 | 76
  >=65 years | 7 | 4 | 11
Age, Continuous [Mean (Standard Deviation); unit: years] | 51.63 (12.36) | 50.38 (13.88) | 51.01 (13.07)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 11 | 13 | 24
  Male | 33 | 30 | 63
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | 0
  Not Hispanic or Latino | 44 | 42 | 86
  Unknown or Not Reported | 0 | 1 | 1
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 1 | 1
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 2 | 1 | 3
  White | 40 | 39 | 79
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 2 | 2 | 4
Region of Enrollment [Number; unit: participants]
  United States | 44 | 43 | 87

OUTCOME MEASURES:

1. Primary Outcome: 6-month Progression-free Survival.
Description: Time between the start of treatment to progression. Progression is defined by the RANO(Response Assessment in Neuro-Oncology) criteria. Progression is defined by any of the following: 25% increase in sum of the products of perpendicular diameters of enhancing lesions; any new lesion; or clinical deterioration.
Time Frame: 6 months
Population: 63 patients enrolled with glioblastoma multiforme (GBM) (32 Bev naive, 31 Bev resistant) and were evaluated for this outcome measure.
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Bevacizumab Resistant Patients | Bevacizumab Naive Patients
Number analyzed (Participants) | 31 | 32
Months | 0.92 [0.89 to 0.92] | 1.08 [0.92 to 2.47]

2. Secondary Outcome: Number of Participants With Adverse Events
Description: Here is the number of participants with adverse events. For a detailed list of adverse events, see the adverse event module.
Time Frame: 7/2/08 -12/6/13
Measure: Number; unit: Participants
Arm/Group | Bevacizumab Resistant Patients | Bevacizumab Naive Patients
Number analyzed (Participants) | 44 | 43
Participants | 44 | 43

ADVERSE EVENTS:
Arm/Group | Bevacizumab Resistant Patients | Bevacizumab Naive Patients
Serious Adverse Events (participants affected / at risk) | 16/44 | 13/43
Other Adverse Events (participants affected / at risk) | 44/44 | 43/43
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Bevacizumab Resistant Patients (N=44) | Bevacizumab Naive Patients (N=43)
Diarrhea (Gastrointestinal disorders) | 1 (1) | 0 (0)
Death not associated with CTCAE term: Death NOS (General disorders) | 1 (1) | 1 (1)
Death not associated with CTCAE term: Disease progression NOS (General disorders) | 4 (4) | 2 (2)
Encephalopathy (Nervous system disorders) | 0 (0) | 1 (1)
Fatigue (asthenia, lethargy, malaise) (General disorders) | 1 (1) | 1 (1)
Gastrointestinal-Other (hemorrhoids) (Gastrointestinal disorders) | 0 (0) | 1 (1)
Infection with normal ANC or Grade 1 or 2 neutrophils::Lung (pneumonia) (Infections and infestations) | 0 (0) | 2 (2)
Pain: Head/Headache (Nervous system disorders) | 1 (1) | 2 (3)
Seizure (Nervous system disorders) | 3 (3) | 1 (1)
Speech impairment (e.g. dysphasia or aphasia) (Nervous system disorders) | 0 (0) | 1 (1)
Supraventricular & nodal arrhythmia: Sinus tachycardia (Nervous system disorders) | 0 (0) | 1 (1)
Thrombosis/thrombus/embolism (Vascular disorders) | 1 (1) | 4 (4)
Cholecystitis (Hepatobiliary disorders) | 1 (1) | 0 (0)
Dehydration (Gastrointestinal disorders) | 1 (1) | 0 (0)
Dizziness (Nervous system disorders) | 1 (1) | 0 (0)
Hemorrhage, CNS (Blood and lymphatic system disorders) | 2 (2) | 0 (0)
Hemorrhage, pulmonary/upper respiratory: Nose (Blood and lymphatic system disorders) | 1 (1) | 0 (0)
Hypertension (Cardiac disorders) | 2 (2) | 0 (0)
Hypotension (Cardiac disorders) | 1 (1) | 0 (0)
Infection (Infections and infestations) | 2 (2) | 0 (0) — (documented clinically or microbiologically) with Grade 3 or 4 neutrophils (ANC <1.0 x 10e9/L): Lung (pneumonia)
Leukocytes (total WBC) (Blood and lymphatic system disorders) | 2 (3) | 0 (0)
Muscle weakness, generalized or specific area (not due to neuropathy): Extremity-upper (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Nausea (Gastrointestinal disorders) | 2 (2) | 0 (0)
Neurology - other (herniation) (Nervous system disorders) | 1 (1) | 0 (0)
Neutrophils/granulocytes (ANC/AGC) (Blood and lymphatic system disorders) | 2 (3) | 0 (0)
Opportunistic infection associated with >=Grade 2 lymphopenia (Infections and infestations) | 1 (1) | 0 (0)
Pancreatitis (Hepatobiliary disorders) | 1 (2) | 0 (0)
Pyramidal tract dysfunction (Nervous system disorders) | 1 (1) | 0 (0) — (e.g. increased tone, hyperflexia, positive Babinski, decreased fine motor coordination)
Vomiting (Gastrointestinal disorders) | 3 (3) | 0 (0)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Bevacizumab Resistant Patients (N=44) | Bevacizumab Naive Patients (N=43)
Diarrhea (Gastrointestinal disorders) | 13 (14) | 7 (11)
Hypertension (Cardiac disorders) | 24 (25) | 13 (18)
ALT/SGPT (serum glutamic pyruvic transaminase) (Metabolism and nutrition disorders) | 21 (25) | 21 (30)
AST/SGOT (serum glutamic oxaloacetic transaminase) (Metabolism and nutrition disorders) | 12 (16) | 10 (10)
Albumin, serum-low (hypoalbuminemia) (Metabolism and nutrition disorders) | 20 (23) | 19 (24)
Alkaline phosphatase (Metabolism and nutrition disorders) | 5 (5) | 6 (6)
Bilirubin (hyperbilirubinemia) (Metabolism and nutrition disorders) | 8 (10) | 9 (10)
CPK (creatine phosphokinase) (Metabolism and nutrition disorders) | 1 (1) | 4 (4)
Cardiac General - Other (mitral valve disease) (Cardiac disorders) | 0 (0) | 1 (1)
Cardiac troponin T (cTnT) (Cardiac disorders) | 0 (0) | 1 (1)
Cognitive disturbance (Nervous system disorders) | 1 (1) | 2 (2)
Constipation (Gastrointestinal disorders) | 2 (2) | 5 (5)
Cough (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Creatinine (Metabolism and nutrition disorders) | 6 (8) | 1 (1)
Cushingoid appearance (e.g. moon face, buffalo hump, centripetal obesity, cutaneous striae) (Endocrine disorders) | 0 (0) | 1 (1)
Dermatology/Skin-Other (skin tear) (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Dyspnea (shortness of breath) (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (1)
Edema: limb (Musculoskeletal and connective tissue disorders) | 1 (1) | 1 (1)
Extremity-lower (gait/walking) (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Fatigue (asthenia, lethargy, malaise) (General disorders) | 8 (9) | 11 (11)
Fever (in the absence of neutropenia, where neutropenia is defined as ANC <1.0 x 10e9/L) (General disorders) | 0 (0) | 2 (3)
Fracture (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Gastrointestinal-Other (tongue irritation, soreness) (Gastrointestinal disorders) | 0 (0) | 1 (1)
Glucose, serum-high (hyperglycemia) (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Glucose, serum-high (hypoglycemia) (Metabolism and nutrition disorders) | 1 (1) | 4 (5)
Heartburn/Dyspepsia (Gastrointestinal disorders) | 4 (4) | 5 (5)
Hemoglobin (Blood and lymphatic system disorders) | 11 (15) | 15 (21)
Hemorrhage, CNS (Blood and lymphatic system disorders) | 1 (1) | 1 (1)
Hemorrhage, GI: Anus (Blood and lymphatic system disorders) | 0 (0) | 2 (2)
Hemorrhage, GI: oral cavity (Blood and lymphatic system disorders) | 0 (0) | 1 (1)
Hemorrhage, pulmonary/upper respiratory: Nose (Blood and lymphatic system disorders) | 3 (3) | 3 (3)
Hiccoughs (hiccups, singultus) (Respiratory, thoracic and mediastinal disorders) | 1 (2) | 1 (1)
Hypopigmentation (Skin and subcutaneous tissue disorders) | 1 (1) | 6 (6)
Hypotension (Cardiac disorders) | 0 (0) | 2 (2)
Infection with normal ANC or Grade 1 or 2 neutrophils::Bronchus (Infections and infestations) | 0 (0) | 1 (1)
Infection with normal ANC or Grade 1 or 2 neutrophils::Lip/perioral (Infections and infestations) | 1 (1) | 1 (1)
Infection with normal ANC or Grade 1 or 2 neutrophils::Upper airway NOS (Infections and infestations) | 1 (1) | 2 (2)
Infection with unknown ANC: Lung (pneumonia) (Infections and infestations) | 1 (1) | 1 (1)
Insomnia (General disorders) | 3 (3) | 3 (3)
Left ventricular diastolic dysfunction (Cardiac disorders) | 0 (0) | 1 (1)
Leukocytes (total WBC) (Blood and lymphatic system disorders) | 25 (40) | 37 (85)
Libido (Reproductive system and breast disorders) | 0 (0) | 1 (1)
Lymphopenia (Blood and lymphatic system disorders) | 24 (35) | 24 (64)
Magnesium, serum-high (hypermagnesemia) (Metabolism and nutrition disorders) | 7 (8) | 6 (6)
Magnesium, serum-low (hypomagnesemia) (Metabolism and nutrition disorders) | 0 (0) | 2 (2)
Metabolic/Laboratory - Other (Elevated LDH; lactate dehidrogenase) (Metabolism and nutrition disorders) | 0 (0) | 2 (2)
Mood alteration: agitation (Nervous system disorders) | 0 (0) | 1 (1)
Mood alteration: depression (Nervous system disorders) | 3 (3) | 1 (1)
Mucositis/stomatitis (clinical exam)::oral cavity (Gastrointestinal disorders) | 2 (2) | 2 (2)
Mucositis/stomatitis (functional/symptomatic)::oral cavity (Gastrointestinal disorders) | 0 (0) | 3 (3)
Muscle weakness, generalized or specific area (not due to neuropathy): Extremity-lower (Musculoskeletal and connective tissue disorders) | 2 (2) | 5 (5)
Muscle weakness, generalized or specific area (not due to neuropathy): Left-sided (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Muscle weakness, generalized or specific area (not due to neuropathy): Right-sided (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Nail changes (Skin and subcutaneous tissue disorders) | 0 (0) | 2 (2)
Nausea (Gastrointestinal disorders) | 3 (4) | 7 (7)
Neurology - Other (decreased concentration; spatial disorientation) (Nervous system disorders) | 0 (0) | 2 (2)
Neuropathy:sensory (Nervous system disorders) | 0 (0) | 1 (1)
Neutrophils/granulocytes (ANC/AGC) (Blood and lymphatic system disorders) | 16 (23) | 27 (51)
Ocular/Visual-Other, color contrast changes; color vision distortion; eisodic wavy vision (Eye disorders) | 0 (0) | 0 (0)
Opportunistic infection associated with >=Grade 2 lymphopenia (Infections and infestations) | 4 (4) | 5 (6)
Pain: Head/Headache (Nervous system disorders) | 6 (6) | 6 (6)
Pain: Joint (Musculoskeletal and connective tissue disorders) | 1 (1) | 4 (5)
Pain: Pain NOS (General disorders) | 0 (0) | 1 (1)
Pain: Throat/pharynx/larynx (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Phosphate, serum-low (hypophosphatemia) (Metabolism and nutrition disorders) | 18 (24) | 17 (24)
Platelets (Blood and lymphatic system disorders) | 30 (52) | 31 (54)
Potassium, serum-high (hyperkalemia) (Metabolism and nutrition disorders) | 3 (3) | 4 (5)
Potassium, serum-low (hypokalemia) (Metabolism and nutrition disorders) | 2 (3) | 2 (2)
Prolonged QTc interval (Cardiac disorders) | 0 (0) | 1 (1)
Proteinuria (Metabolism and nutrition disorders) | 2 (2) | 2 (2)
Pulmonary/Upper respiratory - Other (right upper lobe cavity mass) (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Pyramidal tract dysfunction (Nervous system disorders) | 10 (11) | 2 (2) — (e.g. increased tone, hyperflexia, positive Babinski, decreased fine motor coordination)
Rash/Desquamation (Skin and subcutaneous tissue disorders) | 2 (2) | 8 (8)
Rash: acne/acneiform (Skin and subcutaneous tissue disorders) | 1 (1) | 2 (2)
Rash: erythema multiforme (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) — e.g. Stevens-Johnson syndrome, toxic epidermal necrolysis)
Rash: hand-foot skin reaction (Skin and subcutaneous tissue disorders) | 1 (1) | 1 (1)
Seizure (Nervous system disorders) | 8 (9) | 4 (4)
Sodium, serum-high (hypernatremia) (Metabolism and nutrition disorders) | 0 (0) | 3 (3)
Sodium, serum-low (hyponatremia) (Metabolism and nutrition disorders) | 7 (8) | 4 (5)
Speech impairment (e.g. dysphasia or aphasia) (Nervous system disorders) | 1 (1) | 1 (1)
Supraventricular & nodal arrhythmia: Sinus bradycardia (Cardiac disorders) | 0 (0) | 1 (1)
Taste alteration (dysgeusia) (Gastrointestinal disorders) | 0 (0) | 7 (7)
Thrombosis/thrombus/embolism (Vascular disorders) | 0 (0) | 1 (1)
Thyroid function, high (hyperthyroidism, thyrotoxicosis) (Endocrine disorders) | 1 (1) | 6 (6)
Thyroid function, low (hypothyroidism) (Endocrine disorders) | 20 (20) | 17 (18)
Ulceration (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Vision-blurred vision (Eye disorders) | 0 (0) | 1 (1)
Vomiting (Gastrointestinal disorders) | 0 (0) | 1 (1)
Weight loss (General disorders) | 0 (0) | 1 (1)
Arthritis (non-septic) (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Edema: head and neck (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Memory impairment (Nervous system disorders) | 2 (2) | 0 (0)
Pain: chest wall (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Infection with normal ANC or Grade 1 or 2 neutrophils::Mucosa (Infections and infestations) | 1 (1) | 0 (0)
Skin breakdown/decubitus ulcer (Skin and subcutaneous tissue disorders) | 3 (3) | 0 (0)
Voice changes/dysarthia (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) — (e.g., hoarseness, loss of alteration in voice, laryngitis)
Vision-flashing lights/floaters (Eye disorders) | 2 (2) | 0 (0)
Infection (Infections and infestations) | 1 (1) | 0 (0) — (documented clinically or microbiologically) with Grade 3 or 4 neutrophils (ANC <1.0 x 10e9/L): pancreas
Incontinence, urinary (Renal and urinary disorders) | 3 (3) | 0 (0)
Dizziness (Nervous system disorders) | 1 (1) | 1 (1)
Muscle weakness, generalized or specific area (not due to neuropathy): whole body/generalized (Musculoskeletal and connective tissue disorders) | 0 (0) | 2 (2)
Ataxia (incoordination) (Nervous system disorders) | 1 (1) | 0 (0)
Bruising (in absence of Grade 3 or 4 thrombocytopenia) (Skin and subcutaneous tissue disorders) | 2 (2) | 0 (0)
Confusion (Nervous system disorders) | 3 (3) | 0 (0)
Mood alteration: anxiety (Nervous system disorders) | 2 (2) | 0 (0)
Neurology Other (quadrantanopsia; sensory loss) (Nervous system disorders) | 2 (2) | 0 (0)
Pain: back (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Pain: neck (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Pain: oral cavity (Gastrointestinal disorders) | 1 (1) | 0 (0)
Dermatology/Skin-Other (hair pigmentation changes) (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Ocular/Visual - Other (color contrast changes, color vision distortion, eisodic wavy vision) (Eye disorders) | 0 (0) | 3 (3)
Calcium, serum-low (hypocalcemia) (Metabolism and nutrition disorders) | 3 (3) | 0 (0)
Metabolic/Laboratory - Other (high LDH) (Metabolism and nutrition disorders) | 1 (1) | 0 (0)

LIMITATIONS AND CAVEATS:
The study was terminated based on results of an interim analysis for futility.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No